CLINICAL TRIAL: NCT00137085
Title: Ketamine Versus Fentanyl as an Adjunct to Propofol-Assisted Emergency Department Procedural Sedation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Queen's University (Other)
Collaborators: The Physicians' Services Incorporated Foundation (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: PSI R04-43
Record Dates: First submitted 2005-08-26; First posted 2005-08-29 (Estimated); Last update posted 2007-06-14 (Estimated); Status verified 2006-04

CONDITIONS: Fractures; Dislocations; Abscess; Anesthesia; Analgesia
Keywords: procedural sedation
MeSH Terms: conditions — Fractures, Bone; Joint Dislocations; Abscess; Agnosia | interventions — Ketamine

INTERVENTIONS:
Drug: ketamine

SUMMARY:
We, the investigators at Queen's University, propose to conduct a randomized, double-blind, feasibility trial comparing low-dose ketamine versus fentanyl as adjuncts to Emergency Department procedural sedation with propofol. The outcomes of interest will be safety, with respect to hemodynamic and respiratory adverse effects, as well as efficacy, with respect to adequacy of sedation and analgesia, recovery profiles and patient/physician satisfaction. Our hypothesis, based on a review of existing anesthesia literature, is that low-dose ketamine may be a safer and more efficacious alternative to fentanyl when used as an adjunct to propofol-assisted procedural sedation.

DETAILED DESCRIPTION:
This initial, single-centre feasibility study will have the following specific objectives:

* Comparison of low-dose ketamine with fentanyl as adjunct to propofol-assisted emergency department procedural sedation, with respect to safety and efficacy parameters;
* Pilot of a blinded emergency department sedation and analgesia protocol, including drug doses, concealment techniques, and data collection tools, to determine the feasibility of a subsequent larger, multi-centre trial;
* Determination of the true incidence of the primary outcome measures in the study population, using the study drug administration doses and protocol, such that an accurate sample size may be estimated for a future, adequately-powered, multi-centre trial;
* Validation of a newly-developed ordered, categorical rating scale for the reporting of respiratory and hemodynamic adverse events occurring during emergency department procedural sedation and analgesia.

ELIGIBILITY:
Inclusion Criteria:

* Individuals presenting or referred to the Emergency Department at Kingston General Hospital with a fracture or dislocation requiring manipulation under procedural sedation; or abscess requiring incision and drainage under procedural sedation.
* Ability to provide informed consent according to institutional requirements.
* Ability to comprehend and communicate in English.

Exclusion Criteria:

* Age < 14 or > 65 years
* Any history of significant active cardiac, pulmonary, hepatic or renal disease, as determined by patient history, chart review, or emergency physician.
* American Society of Anesthesiology (ASA) classification greater than class II.
* Body mass > 130 kg.
* A history of physician-diagnosed obstructive sleep apnea.
* Chronic use of opioids including methadone and buprenorphine.
* A self-reported history of recent substance abuse or prior opioid dependence.
* Acute intoxication with drugs or alcohol, based on the judgement of the attending physician.
* A history of psychotic disorders, as reported by subjects or identified on review of the medical records.
* A known history of allergy or sensitivity to any study medication.

Ages: 14 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 124
Dates: Start 2004-09; Study Completion 2006-08 (Actual)

PRIMARY OUTCOMES:
The primary outcome of interest in this study will be the incidence and severity of adverse events during procedural sedation, characterized by using an ordered, four-point categorical scale of airway, ventilatory and hemodynamic adverse events.

SECONDARY OUTCOMES:
The secondary outcome measures of this study will be: the incidence and type of individual adverse events listed in the primary outcome
the dose of propofol administered during the procedure
times from study drug administration to: beginning of procedure, end of procedure, recovery of appropriate verbal response, Emergency Department discharge, incidence of any adverse event(s)
successful completion of the procedure
the operator's rating of the sedation
incidence of any adverse drug reaction
patient visual analogue scale (VAS) ratings of analgesia, amnesia, and general satisfaction.

CONTACTS AND LOCATIONS:
Overall Officials: Marco LA Sivilotti, MD, MSc, Principal Investigator — Queen's University
Locations (1):
- Queen's University, Kingston, Ontario, Canada

REFERENCES:
- [Derived] Messenger DW, Murray HE, Dungey PE, van Vlymen J, Sivilotti ML. Subdissociative-dose ketamine versus fentanyl for analgesia during propofol procedural sedation: a randomized clinical trial. Acad Emerg Med. 2008 Oct;15(10):877-86. doi: 10.1111/j.1553-2712.2008.00219.x. Epub 2008 Aug 27. PMID 18754820